CLINICAL TRIAL: NCT01741532
Title: A Randomized, Double-blind, Placebo-controlled Trial of Deferiprone in Patients With Pantothenate Kinase-associated Neurodegeneration (PKAN)
Brief Title: Efficacy and Safety Study of Deferiprone in Patients With Pantothenate Kinase-associated Neurodegeneration (PKAN)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ApoPharma (Industry)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TIRCON2012V1; 1R01FD004103-01 (FDA)
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Results first posted 2019-05-23 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Pantothenate Kinase-Associated Neurodegeneration
Keywords: Pantothenate Kinase-associated Neurodegeneration; PKAN; NBIA; Deferiprone; Ferriprox; Neurodegeneration with brain iron accumulation
MeSH Terms: conditions — Pantothenate Kinase-Associated Neurodegeneration | interventions — Deferiprone; Isoflurophate; Long Interspersed Nucleotide Elements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo solution matched deferiprone oral solution in appearance, taste, and packaging
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deferiprone (Experimental): Deferiprone 80 mg/mL oral solution
  Interventions: Drug: Deferiprone oral solution
- Placebo (Placebo Comparator): Matching placebo solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Deferiprone oral solution — Deferiprone 80 mg/mL oral solution will be administered twice daily (b.i.d.) for 18 months. An initial dose of 5 mg/kg b.i.d. will be administered for 6 weeks. The dose will then be escalated to 10 mg/kg b.i.d. and finally to 15 mg/kg b.i.d.
  Other Names: DFP; L1
  Arms: Deferiprone
Drug: Placebo — A deferiprone matching placebo oral solution will be given twice daily for 18 months.
  Arms: Placebo

SUMMARY:
A multi-center, placebo controlled, double-blind trial comparing the efficacy and safety of 18 months of treatment with deferiprone versus placebo in patients with PKAN.

This investigator-initiated trial was funded by the European Commission's Seventh Framework Programme (FP7/2007-2013, HEALTH-F2-2011, grant agreement No. 277984) to the TIRCON consortium (Treat Iron-Related Childhood-Onset Neurodegeneration) and by the FDA Office of Orphan Products Development (OOPD) (Dr. Elliott Vichinsky).

DETAILED DESCRIPTION:
This is a multi-center, double-blind, randomized, placebo-controlled, 18-month study in patients with PKAN aged 4 years and older. Participants are randomized in a 2:1 ratio to receive either deferiprone oral solution or placebo, twice a day for 18 months. Efficacy assessments, an MRI scan to measure iron levels in the globus pallidus, pharmacokinetic evaluations, and safety assessments are conducted at specified time points. Following completion of the trial, eligible patients are invited to enroll in an 18-month extension study, TIRCON2012V1-EXT, in which all participants receive deferiprone.

ELIGIBILITY:
Main Inclusion Criteria:

* Males or females 4 years of age and older at screening visit;
* Have PKAN, confirmed by genetic testing (supporting evidence required);
* Barry-Albright Dystonia (BAD) total score ≥ 3 at the screening visit;
* Patients who have Deep Brain Stimulation (DBS) systems or baclofen pumps in place will be eligible for the study, but they must have had a stable setting for at least two months prior to the screening visit and stimulation parameters / pump settings must remain stable for the duration of the trial:

Main Exclusion Criteria:

* Evidence of iron deficiency defined by Fe:TIBC ratio <15%, or serum ferritin <12 ng/mL;
* Treatment with deferiprone in the past 12 months;
* Previous failure of treatment with deferiprone, or previous discontinuation of treatment with deferiprone due to adverse events;
* Conditions known to contraindicate the use of deferiprone (history of agranulocytosis or recurrent episodes of neutropenia);
* A serious, unstable chronic illness not related to PKAN condition during the past 3 months before screening visit including but not limited to: hepatic, renal, gastro-enterologic, respiratory, cardiovascular, endocrinologic, neurologic or immunologic disease;
* Evidence of abnormal liver or renal function (serum liver enzyme level(s) > 3 times upper limit of normal at screening) or abnormal creatinine levels at screening visit;
* Disorders associated with neutropenia (ANC < 1.5 x 10^9/L) or thrombocytopenia (platelet count < 50 x 10^9/L) in the 12 months preceding the initiation of the study medication. Exception: for patients whose neutropenia was attributed by the treating physician to episodes of infection or to drugs associated with a decline in the neutrophil count and in whom the ANC has fully recovered at the screening visit;
* History of malignancy;

Other protocol inclusion or exclusion criteria may apply.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2012-12-13 (Actual); Primary Completion 2016-10-21 (Actual); Study Completion 2017-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Tricta, MD, Study Chair — ApoPharma Inc.; Thomas Klopstock, MD, Principal Investigator — Friedrich-Baur-Institute, Department of Neurology, University of Munich Ziemssenstr; Elliott Vichinsky, MD, Principal Investigator — Children's Hospital & Research Center at Oakland Hematology/ Oncology, Pediatric Rehabilitation
Locations (4):
- Children's Hospital & Research Center at Oakland, Oakland, California, United States
- Klinikum der Universität München, Munich, Germany
- Foundation Neurological Institute C. Besta, Milan, Italy
- Newcastle University Institute of Human Genetics, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Derived] Klopstock T, Tricta F, Neumayr L, Karin I, Zorzi G, Fradette C, Kmiec T, Buchner B, Steele HE, Horvath R, Chinnery PF, Basu A, Kupper C, Neuhofer C, Kalman B, Dusek P, Yapici Z, Wilson I, Zhao F, Zibordi F, Nardocci N, Aguilar C, Hayflick SJ, Spino M, Blamire AM, Hogarth P, Vichinsky E. Safety and efficacy of deferiprone for pantothenate kinase-associated neurodegeneration: a randomised, double-blind, controlled trial and an open-label extension study. Lancet Neurol. 2019 Jul;18(7):631-642. doi: 10.1016/S1474-4422(19)30142-5. PMID 31202468

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 4 study sites in Germany, Italy, the U.K., and the U.S.
Groups:
- Deferiprone: Patients randomized to this arm received deferiprone oral solution 80 mg/mL at a dosage of up to 15 mg/kg twice a day for up 18 months.
- Placebo: Patients randomized to this arm received matching placebo solution twice a day, for up to 18 months, at a volume corresponding to that taken by patients who were receiving active product.
Period: Overall Study
Arm/Group | Deferiprone | Placebo
Started | 59 | 30
Exposed | 58 | 30
Provided Post-baseline Efficacy Data | 58 | 28
Completed | 49 | 27
Not Completed | 10 | 3
Not completed — Adverse Event | 4 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Worsening of the disease | 3 | 1
Not completed — Sponsor decision | 1 | 0
Not completed — Medical event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Deferiprone: Deferiprone 80 mg/mL oral solution, 15 mg/kg b.i.d. for 18 months
- Placebo: Matching volume of placebo solution, twice daily for 18 months
- Total: Total of all reporting groups
Arm/Group | Deferiprone | Placebo | Total
Number analyzed (Participants) | 59 | 30 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.8 (10.7) | 19.2 (12.5) | 20.2 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 17 | 42
  Male | 34 | 13 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 51 | 28 | 79
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Score on Barry-Albright Dystonia Scale
Description: The Barry-Albright Dystonia (BAD) scale rates severity of dystonia (sustained muscle contractions causing twisting and repetitive movements or abnormal postures) in 8 body regions. The individual scores are summed to provide a total score ranging from 0 to 32, with higher scores indicating greater severity. The co-primary endpoint in this study was the change from baseline to Month 18 in BAD total score.
Time Frame: Baseline to 18 Months
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Deferiprone: Patients randomized to this arm received deferiprone oral solution 80 mg/mL at a dosage of up to 15 mg/kg twice a day for up to 18 months.
- Placebo: Patients randomized to this arm received matching placebo solution twice a day, for up to 18 months, at a volume corresponding to what was given for the active product.
Arm/Group | Deferiprone | Placebo
Number analyzed (Participants) | 58 | 28
score on a scale | 2.48 (0.63) | 3.99 (0.82)
Statistical Analysis 1: Comparison: Deferiprone vs Placebo; Test type: Superiority; p = 0.0761, Mixed Models Analysis

2. Primary Outcome: Score on Patient Global Impression of Improvement at End of Study
Description: The Patient Global Impression of Improvement (PGI-I) is a global index that assesses the response of a condition to a therapy by asking patients to rate their current state relative to their state at baseline. It consists of a 7-point rating scale, where 1=very much improved, 2= much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse.
Time Frame: Month 18
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Deferiprone | Placebo
Number analyzed (Participants) | 58 | 28
score on a scale | 4.55 (0.30) | 4.66 (0.38)
Statistical Analysis 1: Comparison: Deferiprone vs Placebo; Test type: Superiority; p = 0.7279, Mixed Models Analysis

3. Secondary Outcome: Change in Score on Unified Parkinson's Disease Rating Scale
Description: The Unified Parkinson's Disease Rating Scale (UPDRS) is the major rating scale used to assess severity of symptoms of Parkinson's disease, some of which are similar to those of PKAN. The UPDRS subscales used in this study were Part I: Mentation, Behavior and Mood, scored from 0 (best) to 16 (worst); Part II: Activities of Daily Living, scored from 0 (best) to 52 (worst); Part III: Motor Examination, scored from 0 (best) to 108 (worst); and Part VI: Schwab and England Activities of Daily Living Scale, scored from 0% (worst) to 100% (best).
Time Frame: Baseline to 18 Months
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Deferiprone | Placebo
Number analyzed (Participants) | 58 | 28
score on a scale
  UPDRS Part I | -0.25 (0.43) | -0.07 (0.55)
  UPDRS Part II | 1.09 (1.19) | 2.36 (1.52)
  UPDRS Part III | 5.38 (2.20) | 2.06 (2.79)
  UPDRS Part VI | -2.17 (2.94) | -7.66 (3.85)
Statistical Analysis 1: Comparison: Deferiprone vs Placebo; Comparison of treatment groups on change in score on UPDRS Part I; Test type: Superiority; p = 0.7228, Mixed Models Analysis
Statistical Analysis 2: Comparison: Deferiprone vs Placebo; Comparison of treatment groups on change in score on UPDRS Part II; Test type: Superiority; p = 0.3677, Mixed Models Analysis
Statistical Analysis 3: Comparison: Deferiprone vs Placebo; Comparison of treatment groups on change in score on UPDRS Part III; Test type: Superiority; p = 0.2182, Mixed Models Analysis
Statistical Analysis 4: Comparison: Deferiprone vs Placebo; Comparison of treatment groups on change in score on UPDRS Part VI; Test type: Superiority; p = 0.1749, Mixed Models Analysis

4. Secondary Outcome: Change in Score on Functional Independence Measure
Description: The Functional Independence Measure (FIM) scale is used to assess physical and cognitive disability in three areas of daily living: self-care, mobility, and cognition. Within each area, items are scored according to the level of assistance required to perform that activity of daily living. A score of 1-2 indicates that the patient is completely dependent on a helper to perform the task, a score of 3-5 indicates that the patient is moderately dependent, and a score of 6-7 indicates that no help is required. The individual scores are summed to provide a global score from 18 (worst) to 126 (best).
Time Frame: Baseline to 18 Months
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Deferiprone | Placebo
Number analyzed (Participants) | 58 | 28
score on a scale | 5.40 (2.36) | 0.69 (3.34)
Statistical Analysis 1: Comparison: Deferiprone vs Placebo; Test type: Superiority; p = 0.1524, Mixed Models Analysis

5. Secondary Outcome: Change in Score on WeeFIM
Description: The WeeFIM is the pediatric version of the Functional Independence Measure scale, and is used to assess physical and cognitive disability in three areas of daily living: self-care, mobility, and cognition. Within each area, items are scored according to the level of assistance required to perform that activity of daily living. A score of 1-2 indicates that the patient is completely dependent on a helper to perform the task, a score of 3-5 indicates that the patient is moderately dependent, and a score of 6-7 indicates that no help is required. The individual scores are summed to provide a global score from 18 (worst) to 126 (best).
Time Frame: Baseline to 18 Months
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Deferiprone | Placebo
Number analyzed (Participants) | 58 | 28
score on a scale | 4.91 (5.30) | -2.40 (5.42)
Statistical Analysis 1: Comparison: Deferiprone vs Placebo; Test type: Superiority; p = 0.2026, Mixed Models Analysis

6. Secondary Outcome: Change in Score on Pediatric Quality of Life
Description: The Pediatric Quality of Life (PedsQL) questionnaire is used to measure functional health and well-being from the patient's point of view. Separate versions of the questionnaire are available for children, young adults aged 18-25 years, and adults older than 25 years. Patients are asked to indicate how they have felt over the past month, and the scores of the 23 questions are used to generate an overall score that ranges from 0 (worst) to 100 (best).
Time Frame: Baseline to 18 Months
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Deferiprone | Placebo
Number analyzed (Participants) | 58 | 28
score on a scale
  Patient self-report, total score | 1.21 (3.68) | 1.34 (4.49)
  Parent proxy-report, total score | -4.90 (3.99) | -2.37 (4.90)
Statistical Analysis 1: Comparison: Deferiprone vs Placebo; Patient self-report, total score; Test type: Superiority; p = 0.9759, Mixed Models Analysis
Statistical Analysis 2: Comparison: Deferiprone vs Placebo; Parent proxy-report, total score; Test type: Superiority; p = 0.5781, Mixed Models Analysis

7. Secondary Outcome: Change in Score on Pittsburgh Sleep Quality Index
Description: The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire that assesses sleep quality and disturbances over a 1-month time interval. A total of 19 individual items are used to generate 7 "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction, and a score is generated that ranges from 0 (best) to 21 (worst).
Time Frame: Baseline to 18 Months
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Deferiprone | Placebo
Number analyzed (Participants) | 58 | 28
score on a scale | 0.48 (0.61) | 0.14 (0.80)
Statistical Analysis 1: Comparison: Deferiprone vs Placebo; Test type: Superiority; p = 0.6323, Mixed Models Analysis

8. Secondary Outcome: Change in Level of Brain Iron
Description: Neurodegeneration in patients with PKAN is associated with localized brain iron accumulation, with the highest amount of accumulation seen in the globus pallidus, one of the main areas for motor control. MRI R2* scans of this region were performed at baseline and Month 18 in a subset of patients who did not have a deep brain stimulation (DBS) device implanted, and for whom the use of anesthesia, if required, was deemed acceptable by the investigator.
Time Frame: Baseline to 18 Months
Measure: Least Squares Mean (Standard Error); unit: Hz
Groups:
- Deferiprone: The subset of deferiprone recipients who underwent MRI R2* imaging
- Placebo: The subset of placebo recipients who underwent MRI R2* imaging
Arm/Group | Deferiprone | Placebo
Number analyzed (Participants) | 24 | 16
Hz | -36.1 (3.11) | -0.50 (3.97)
Statistical Analysis 1: Comparison: Deferiprone vs Placebo; Test type: Superiority; p = 0.0000, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline until 30 days after the last dose of study medication.
Groups:
- Deferiprone: Study participants who received at least one dose of deferiprone in the trial
- Placebo: Study participants who received at least one dose of placebo in the trial
Arm/Group | Deferiprone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/30
Serious Adverse Events (participants affected / at risk) | 18/58 | 10/30
Other Adverse Events (participants affected / at risk) | 57/58 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferiprone (N=58) | Placebo (N=30)
Neutropenia (Blood and lymphatic system disorders) | 5 (7) | 2 (2)
Intestinal dilatation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Condition aggravated (General disorders) | 0 (0) | 1 (1)
Obstruction (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Bacterial disease carrier (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Chemical eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Unintentional medical device removal (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Medical observation (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dystonia (Nervous system disorders) | 3 (3) | 2 (3)
Hypotonia (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Oromandibular dystonia (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Device malfunction (Product Issues) | 1 (1) | 0 (0)
Staring (Psychiatric disorders) | 0 (0) | 1 (1)
Urinary bladder rupture (Renal and urinary disorders) | 1 (1) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Colectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Gastrointestinal tube insertion (Surgical and medical procedures) | 1 (1) | 1 (1)
Intestinal anastomosis (Surgical and medical procedures) | 1 (1) | 0 (0)
Intrathecal pump insertion (Surgical and medical procedures) | 1 (2) | 0 (0)
Laparotomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Medical device battery replacement (Surgical and medical procedures) | 2 (2) | 1 (1)
Nasal septal operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Tracheostomy (Surgical and medical procedures) | 1 (3) | 0 (0)
Tracheostomy tube removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Wound treatment (Surgical and medical procedures) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferiprone (N=58) | Placebo (N=30)
Anaemia (Blood and lymphatic system disorders) | 12 (23) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 2 (3) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 4 (6) | 5 (7)
Constipation (Gastrointestinal disorders) | 2 (3) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 4 (7) | 3 (8)
Influenza (Gastrointestinal disorders) | 3 (4) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 2 (3)
Vomiting (Gastrointestinal disorders) | 9 (17) | 8 (19)
Abasia (General disorders) | 2 (2) | 2 (2)
Condition aggravated (General disorders) | 10 (12) | 9 (10)
Pain (General disorders) | 4 (4) | 0 (0)
Pyrexia (General disorders) | 16 (34) | 13 (28)
Bronchitis (Infections and infestations) | 7 (15) | 2 (2)
Ear infection (Infections and infestations) | 0 (0) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 3 (3) | 3 (4)
Localised infection (Infections and infestations) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 11 (20) | 6 (10)
Rhinitis (Infections and infestations) | 4 (6) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 8 (9) | 4 (5)
Viral infection (Infections and infestations) | 4 (5) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 2 (4)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 6 (15) | 3 (3)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 2 (4)
Blood iron decreased (Investigations) | 3 (3) | 2 (2)
Body temperature increased (Investigations) | 3 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 10 (18) | 3 (20)
Serum ferritin decreased (Investigations) | 19 (23) | 5 (5)
White blood cell count increased (Investigations) | 0 (0) | 2 (2)
Iron deficiency (Metabolism and nutrition disorders) | 9 (9) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (8)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (13) | 4 (7)
Aphasia (Nervous system disorders) | 3 (3) | 2 (2)
Drooling (Nervous system disorders) | 2 (2) | 2 (2)
Dystonia (Nervous system disorders) | 25 (49) | 14 (20)
Freezing phenomenon (Nervous system disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 13 (43) | 9 (30)
Migraine (Nervous system disorders) | 3 (21) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 3 (4) | 2 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 2 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 5 (9)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor retained title to and the right to publish all documentation, records, raw data, specimens or other work product generated in connection with the trial. Such publications shall not be made without the prior written consent of Sponsor. Neither Party will use the other Party's name in connection with any publication or promotion without the other Party's prior written consent. However, Sponsor has the right to publish appropriate information in order to satisfy regulatory requirements.